CLINICAL TRIAL: NCT01631500
Title: Effects of an Integrative Treatment Model to Reduce Anxiety and Depression in Minor Mental Health Problems and Medically Unexplained Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Ekhagastiftelsen (Other); Fyrbodal Research and Development Council (Unknown); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University of Gothenburg; VGFOUREG-82511 (Other Grant/Funding Number: Ekhagastiftelsen 2009-6, RDU Fyrbodal VGFOUFBD-70831)
Record Dates: First submitted 2011-12-08; First posted 2012-06-29 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-06

CONDITIONS: Depression; Anxiety; Irritable Bowel Syndrome; Fibromyalgia
Keywords: Integrative medicine; Acupuncture; Minor mental health problems; Medically unexplained symptoms; Minor mental health problems (e.g. minor depression and anxiety) and Medically unexplained symptoms (e.g. IBS, fibromyalgia, etc)
MeSH Terms: conditions — Depression; Anxiety Disorders; Irritable Bowel Syndrome; Fibromyalgia; Medically Unexplained Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional treatment (Other): Patients receive usual treatments provided at primary care settings, e.g. antidepressants, sessions with a curator or psychotherapist and physiotherapy.
  Interventions: Behavioral: Conventional treatment
- Integrative treatment (Experimental): Person-centred dialogue combined with therapeutic acupuncture (mild manual acupuncture with deqi). Eight individual sessions, once a week, duration approximately 60 minutes
  Interventions: Other: Integrative treatment
- Terapeutic acupuncture (Active Comparator): Therapeutic acupuncture alone, eight individual sessions, once a week. The participants received acupuncture needles in the appropriate acupuncture points, in the same way as the integrative treatment model, but without person-centred dialogue.
  Interventions: Other: Therapeutic acupuncture

INTERVENTIONS:
Behavioral: Conventional treatment — Conventional treatment
  Arms: Conventional treatment
Other: Integrative treatment — Person-centred dialogue combined with therapeutic acupuncture (mild manual acupuncture with deqi). Eight individual sessions, once a week, duration approximately 60 minutes
  Arms: Integrative treatment
Other: Therapeutic acupuncture — Eight individual sessions, once a week, with therapeutic acupuncture. The participants received acupuncture needles in the appropriate acupuncture points, in the same way as the integrative treatment model, but without person-centred dialogue.
  Arms: Terapeutic acupuncture

SUMMARY:
Minor mental health problems, MMHP, like mild depression and anxiety, and medically unexplained symptoms, MUS, symptoms with no known underlying organic disease, are strongly associated to each other. MMHP and MUS have an impact on well-being and quality of life, lead to impaired social and cognitive function and could result in reduced work capacity. The investigators have designed the present study as a pragmatic trial to investigate the effectiveness of an integrative treatment model, therapeutic acupuncture, versus conventional treatment in patients with MMHP or MUS in primary care. The investigators examined whether the effects of the integrative treatment model differed from those achieved with therapeutic acupuncture or conventional treatment. Primary endpoints were anxiety and depression (assessed with the Hospital Anxiety and Depression scale), health-related quality of life (SF-36) and coping with stress, sense of coherence (SOC) during the eight weeks of treatment interventions.

Statistical power was calculated based on an expected 50% reduction in HAD anxiety and depression scores after eight weeks of integrative treatment; a 30% reduction in acupuncture; and 20% in conventional care. A total of 120 (40/arm) were needed to achieve a power of 83% at p <0.05. Treatment effects were calculated as the difference between values at baseline, after four weeks and after the complete intervention period, i.e. after eight weeks. Nonparametric analyses were carried out to test differences between independent samples (Kruskal-Wallis and Mann-Whitney U) and related samples (Wilcoxon).

ELIGIBILITY:
Inclusion Criteria:

* one or more symptoms of emotional and physical fatigue
* worry
* anxiety
* depression
* sleep disturbances or somatic pain

Exclusion Criteria:

* 100% sick leave > 2,5 years
* pregnancy
* cancer
* personality disorders
* substance use disorders or prescribed sedative drugs

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pre-post treatment change in anxiety as assessed with the Hospital Anxiety and Depression scale (HAD) | Baseline and after eight weeks of treatment completion
  Change in HAD Anxiety between baseline and 8-week follow up

SECONDARY OUTCOMES:
Pre-post treatment change in health-related quality of life (assessed with the SF-36 Mental Component Summary score(MCS)) | Baseline and after eight weeks of treatment completion
  Change in SF-36 MCS scores between baseline and 8-week follow up.
Pre-post treatment change in sense of coherence (SOC) | Baseline and after eight weeks of treatment completion
  Change in SOC scores between baseline and 8-week follow up
Pre-post treatment change in depression as assessed with the Hospital Anxiety and Depression scale (HAD) | Baseline and after eight weeks of treatment completion
  Change in HAD Depression scores between baseline and 8-week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Charles Taft, associate professor, Principal Investigator — Göteborg University
Locations (1):
- Fyrbodal Research and Development Council, Vänersborg, Sweden

REFERENCES:
- [Derived] Arvidsdotter T, Marklund B, Taft C, Kylen S. Quality of life, sense of coherence and experiences with three different treatments in patients with psychological distress in primary care: a mixed-methods study. BMC Complement Altern Med. 2015 Apr 26;15:132. doi: 10.1186/s12906-015-0654-z. PMID 25928131
- [Derived] Arvidsdotter T, Marklund B, Taft C. Six-month effects of integrative treatment, therapeutic acupuncture and conventional treatment in alleviating psychological distress in primary care patients--follow up from an open, pragmatic randomized controlled trial. BMC Complement Altern Med. 2014 Jun 30;14:210. doi: 10.1186/1472-6882-14-210. PMID 24980440
- [Derived] Arvidsdotter T, Marklund B, Taft C. Effects of an integrative treatment, therapeutic acupuncture and conventional treatment in alleviating psychological distress in primary care patients--a pragmatic randomized controlled trial. BMC Complement Altern Med. 2013 Nov 7;13:308. doi: 10.1186/1472-6882-13-308. PMID 24200100